CLINICAL TRIAL: NCT00552149
Title: A Multicenter, Randomized Phase II Trial Assessing the Activity of Gemcitabine - Oxaliplatin Chemotherapy Alone or in Combination With Cetuximab in Patients With Advanced Biliary Cancer.
Brief Title: Biliary Cancers: EGFR INhibitor, Gemcitabine and Oxaliplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BINGO; CSET 1287
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2007-10

CONDITIONS: Advanced Biliary Cancer
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): GEMOX
  Interventions: Drug: Gemox, Cetuximab
- 2 (Experimental): GEMOX + CETUXIMAB
  Interventions: Drug: Gemox, Cetuximab

INTERVENTIONS:
Drug: Gemox, Cetuximab — GEMOX (Arms 1 and 2), every two weeks:
  Day 1: gemcitabine 1000 mg/m² intravenous (IV) infusion over 100 minutes (10 mg/m²/min) Day 2: oxaliplatin 100 mg/m² IV infusion over 2 h
  Cetuximab (ErbituxÒ) (Arm B only) every two weeks:
  (chemotherapy will be started one hour after the end of the cetuximab infusion).
  Day 1 or Day 2: 500 mg/m² IV infusion over 150 minutes

SUMMARY:
A Multicenter, Randomized Phase II Trial Assessing the Activity of Gemcitabine - Oxaliplatin Chemotherapy Alone or in Combination with Cetuximab in Patients with Advanced Biliary Cancer.

DETAILED DESCRIPTION:
The BINGO trial is an open-label randomized phase II study evaluating the efficacy and tolerance of gemcitabine-oxaliplatin combination chemotherapy (GEMOX regimen) alone or in combination with cetuximab in patients (pts) with ABC. The BINGO study also comprises ancillary translational research and functional imaging studies which aim to identify markers predictive for treatment efficacy in ABC.

All eligible pts will be randomized 1:1 to receive:

* Arm A: GEMOX alone every two weeks.
* Arm B: GEMOX + cetuximab every two weeks.

Randomization will be stratified according to:

1. tumor stage (locally advanced vs metastatic),
2. primary tumor location (gallbladder vs non-gallbladder),
3. prior treatments (surgery or radiotherapy or brachytherapy or photodynamic therapy [PDT] or adjuvant chemotherapy vs none),
4. center. EGFR tumor status has to be assessed for every pt by immunohistochemistry (IHC) using biopsy or surgical material, at any time prior to inclusion into the study, but it is neither an inclusion/exclusion criterion nor a stratification factor.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the biliary tract (gallbladder, intra and/or extrahepatic bile ducts, or ampulla of Vater):

   * Cytologically or histologically confirmed. In case of uncertain biliary tract origin (e.g., intrahepatic, peripheral cholangiocarcinomas), inclusion is possible if i) extensive search for primary (thoracic and abdominopelvic CT scan, colonoscopy, upper digestive endoscopy, serum PSA level for men or mammography for women, and FDG-PET if possible) is negative; and ii) histological examination is consistent with bile duct adenocarcinoma (IHC should ideally be performed and be consistent with biliary primary, e.g., positive for cytokeratin 7 and 19 and negative for cytokeratin 20).
   * not amenable to curative resection, or recurrent after resection (i.e., locally advanced or metastatic),
   * With at least one unidimensionally measurable target lesion in a non-irradiated, non-PDT-treated area (longest diameter 1 cm [spiral CT scan]), or 2 cm [conventional CT scan]).
   * With biliary obstruction controlled,
2. Age between 18 and 75 years.
3. World Health Organization (WHO) performance status of 0 or 1.
4. Life expectancy higher than 3 months.
5. No prior chemotherapy for advanced disease. Previous adjuvant chemotherapy is allowed (completed at least 6 months previously, if containing gemcitabine or platinum salts). Previous irradiation (external radiotherapy, brachytherapy) and PDT are allowed provided that there is at least one unidimensionally measurable target lesion in untreated area.
6. Bilirubin 3 times the upper limit of the normal range (ULN). Pts with jaundice or evidence of bile duct obstruction, in whom the biliary tree can be decompressed by endoscopic or percutaneous endoprothesis with subsequent reduction in bilirubin £ 3 ULN, will be eligible for the study.
7. Aminotransferases (AST, ALT) 5 ULN, INR < 1.5 (following vitamin K1 injection in patients with current or recent history of jaundice or bile duct obstruction), creatinine 1.5 ULN, neutrophils 1.5 109/L, platelets 100 109/L, hemoglobin 9 g/dL (red blood cell transfusion if needed is allowed).
8. Written informed consent. Note: EGFR tumor status has to be known for every pt, but it is neither an inclusion/exclusion criterion nor a stratification factor. EGFR expression has to be assessed by IHC using biopsy or surgical material, at any time prior to inclusion into the study.

Exclusion Criteria:

1. Known central nervous system metastases.
2. Contraindication or history of grade 3-4 allergy reaction to one treatment component.
3. Surgery (except diagnostic biopsy), external radiotherapy, brachytherapy, or PDT within 30 days prior to start of treatment. Prior adjuvant chemotherapy is only allowed if completed at least 30 days previously (6 months if containing gemcitabine or platinum salts).
4. Participation in another clinical trial within 30 days prior to start of treatment.
5. Concomitant systemic chronic immunotherapy, chemotherapy, or antitumor hormone therapy.
6. Previous administration of EGFR inhibitors or EGF.
7. Active uncontrolled infection, peripheral neuropathy grade 2, acute or subacute bowel obstruction or history of inflammatory bowel disease, symptomatic coronary disease or myocardial infarction in the past 6 months, congestive heart failure (NYHA class II), interstitial pneumonitis or respiratory failure, or renal failure.
8. Pregnancy (or positive b-HCG dosage at baseline), breast-feeding, or lack of effective contraception in male or female pts of reproductive potential.
9. Other malignancies either currently active or in the last 5 years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma.
10. Legal incapacity or physical, psychological or mental status interfering with the pt's ability to terminate the study or to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment efficacy by assessing the crude progression-free survival (PFS) rate at 4 months | 4 months

SECONDARY OUTCOMES:
Evaluation of feasibility and toxicity of the treatments | one year
Evaluation of rate and duration of objective tumor response | one year
Evaluation of rate and duration of tumor control (objective responses and stabilizations) | one year
Evaluation of PFS and over | one year

CONTACTS AND LOCATIONS:
Overall Officials: David MALKA, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Malka D, Cervera P, Foulon S, Trarbach T, de la Fouchardiere C, Boucher E, Fartoux L, Faivre S, Blanc JF, Viret F, Assenat E, Seufferlein T, Herrmann T, Grenier J, Hammel P, Dollinger M, Andre T, Hahn P, Heinemann V, Rousseau V, Ducreux M, Pignon JP, Wendum D, Rosmorduc O, Greten TF; BINGO investigators. Gemcitabine and oxaliplatin with or without cetuximab in advanced biliary-tract cancer (BINGO): a randomised, open-label, non-comparative phase 2 trial. Lancet Oncol. 2014 Jul;15(8):819-28. doi: 10.1016/S1470-2045(14)70212-8. Epub 2014 May 19. PMID 24852116